CLINICAL TRIAL: NCT06832124
Title: Modulating Alpha-connectivity in Patients with Active Suicidal Ideation Using Transcranial Alternating Current Stimulation
Brief Title: Personalized TACS to Reduce Rumination in Patients with Active Suicidal Ideation
Acronym: Alpha-MOD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sebastian Olbrich (Other)
Responsible Party: Sponsor-Investigator, Sebastian Olbrich, Prof. Dr. med., University of Zurich
Organization: University of Zurich (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024-02027
Record Dates: First submitted 2025-02-04; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Suicidal Ideation Active; Depression Disorders
Keywords: tACS; Suicidal ideation; Rumination; Entrapment; Depression; Non-invasive brain stimulation; Suicidal thoughts and behavior
MeSH Terms: conditions — Suicidal Ideation; Rumination Syndrome; Depression; Behavior

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Investigators assessing primary electroencephalography (EEG) outcomes will also be blinded to the assigned study arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sham tACS (Sham Comparator): Participants assigned to this arm will receive active stimulation during one of the stimulation visits and sham stimulation for the remaining one. Sham will involve 10s ramp-up with the same stimulation protocol as the active one, followed by an immediate 10s ramp-down (no stimulation afterwards).
  Interventions: Procedure: Sham alpha-tACS
- Active tACS (Experimental): Participants will receive active tACS during all stimulation visits. The stimulation frequency will be adjusted to the individual alpha peak frequency with in-phase stimulation in parieto-occipital brain areas and anti-phase stimulation in frontal brain areas.
  Interventions: Procedure: alpha-tACS

INTERVENTIONS:
Procedure: Sham alpha-tACS — A sinusoidal ± 2mA current adjusted to the individual alpha peak frequency with in-phase stimulation at parieto-occipital brain areas and anti-phase stimulation in frontal brain areas. The stimulation will involve a 10s ramp-up, followed by an immediate 10s ramp-down (no stimulation afterwards).
  Arms: Sham tACS
Procedure: alpha-tACS — Active tACS with a sinusoidal ± 2mA current adjusted to the individual alpha peak frequency with a 10s ramp-up and 10s ramp-down after stimulation. In-phase stimulation will be applied to parieto-occipital brain areas and anti-phase stimulation will be applied to frontal brain areas
  Arms: Active tACS

SUMMARY:
The goal of this clinical trial is to determine whether modulating default mode network (DMN) alpha connectivity using transcranial alternating current stimulation (tACS) can reduce rumination and, in turn, mitigate feelings of entrapment and suicidal ideation in individuals with active suicidal ideation and depression.

The main questions it aims to answer are:

1. Is personalized tACS stimulation of the DMN associated with reduced rumination 24 hours after stimulation?
2. Does a reduction in rumination result in lower feelings of entrapment and suicidal ideation?
3. Does personalized tACS stimulation of the DMN lead to a reduction of DMN alpha connectivity?

Researchers will compare active tACS stimulation to sham stimulation to assess whether modulating alpha connectivity has a specific effect on rumination, entrapment, suicidal ideation, and DMN alpha connectivity.

Participants will:

* Receive either active or sham tACS stimulation during stimulation sessions, but all participants will receive active tACS at least once.
* Complete self-report measures of rumination, entrapment, and suicidal ideation before and after stimulation.
* Undergo EEG recordings to assess changes in DMN alpha connectivity.

This clinical trial will be preceded by a pilot study in healthy participants with an anticipated completion of data collection in August 2025.

ELIGIBILITY:
Inclusion Criteria:

* Active suicidal ideation defined by a score ≥3 on item #10 of the Montgomery-Asberg Depression Rating Scale (MADRS) and a combined score of ≥2 on items #4 + #5 of the Beck Scale for Suicide Ideation (BSS)
* Clinical diagnosis of a mild to severe depressive episode without psychotic symptoms
* Voluntary patients at inpatient, outpatient, or day-clinic units of mental health care settings in the greater Zurich area
* Aged 18-65 years
* Fluent in German
* Ability to give written informed consent

Exclusion Criteria:

* Mental disorders due to known physiological conditions
* Schizophrenia, schizotypal, delusional, and other non-mood psychotic disorders
* Intellectual disabilities
* Concurrent vagus nerve stimulation, transcranial magnetic stimulation, electro-convulsive therapy, or treatment with nitrous oxide
* Pregnancy or breast-feeding
* Chronic migraines
* Metal implants or any other factor that - in the investigators' judgment - would unduly affect patient safety or compliance during this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
EEG alpha functional connectivity (phase synchronization) | Pre-stimulation to post-stimulation at visit 2 (up to 1 hour)
  The primary outcome measure will be changes in EEG alpha functional connectivity between pre- and post-stimulation at visit 2 (stimulation visit 1) in the active versus sham group (between-person comparison).
  EEG alpha functional connectivity will also be assessed at visit 4 (stimulation visit 2). Allowing for between- and within-person comparisons as secondary outcomes.
Response style questionnaire (RSQ-10D) | Visit 2 to visit 3 (24 hours)
  The primary outcome will be changes in rumination between visit 2 (pre-stimulation) and visit 3 (24 hours post-stimulation) in the active versus sham group (between-person comparison).
  Rumination will also be assessed at visit 4 and visit 5, allowing for between- and within-person comparisons as secondary outcome measures.
  The RSQ-10D measures two facets of rumination: brooding and reflection with 5 items each. Scores per facet range from 5 to 20 with higher scores indicating higher rumination.

SECONDARY OUTCOMES:
Beck Scale for Suicide Ideation (BSS) | Visits 2-5 (24 hours)
  Changes in suicidal ideation between pre-stimulation (visit 2 and visit 4) and post-stimulation (visit 3 and visit 5), between- and within-person comparisons.
  The BSS is a 19-item scale measuring suicidal ideation, with two additional items assessing a history of suicide attempts. Scores range from 0 to 38 with higher scores indicating higher severity of suicidal ideation.
Clinical Global Impression of Imminent Suicide Risk (CGI-SR-I) | Visits 2-5 (24 hours)
  Changes in risk for suicide between pre-stimulation (visit 2 and visit 4) and post-stimulation (visit 3 and visit 5), between- and within-person comparisons.
  The CGI-SR-I is a single-item clinician rating scale where 1 indicates "no imminent suicide risk" and 7 indicates "extreme imminent suicide risk"
Clinical Global Impression of Imminent Suicide Risk (CGI-SR-I) | Visits 2 & 4 (up to 1 hour)
  Changes in risk for suicide between pre-stimulation at visit 2 and visit 4 and post-stimulation at visit 2 and visit 4, between- and within-person comparisons.
  The CGI-SR-I is a single-item clinician rating scale where 1 indicates "no imminent suicide risk" and 7 indicates "extreme imminent suicide risk"
Clinical Global Impression of Suicidality (CGI-SS-R) | Visits 2-5 (24 hours)
  Changes in risk for suicide between pre-stimulation (visit 2 and visit 4) and post-stimulation (visit 3 and visit 5), between- and within-person comparisons.
  The CGI-SS-R is a single-item clinician rating scale where 1 indicates "normal, not at all suicidal" and 7 indicates "among the most extremely suicidal patients"
Clinical Global Impression of Suicidality (CGI-SS-R) | Visits 2 & 4 (up to 1 hour)
  Changes in risk for suicide between pre-stimulation at visit 2 and visit 4 and post-stimulation at visit 2 and visit 4, between- and within-person comparisons.
  The CGI-SS-R is a single-item clinician rating scale where 1 indicates "normal, not at all suicidal" and 7 indicates "among the most extremely suicidal patients"
Suicidal Intent Visual Analogue Scale (S-VAS) | Visits 2-5 (24 hours)
  Changes in suicidal intent between pre-stimulation (visit 2 and visit 4) and post-stimulation (visit 3 and visit 5), between- and within-person comparisons.
  The S-VAS is a single-item visual analogue scale. Scores range from 0 to 100 with 0 indicating "no urge to kill myself" and 100 indicating "extreme urge to kill myself"
Suicidal Intent Visual Analogue Scale (S-VAS) | Visits 2 & 4 (up to 1 hour)
  Changes in suicidal intent between pre-stimulation at visit 2 and visit 4 and post-stimulation at visit 2 and visit 4, between- and within-person comparisons.
  Scores range from 0 to 100 with 0 indicating "no urge to kill myself" and 100 indicating "extreme urge to kill myself".
Short Defeat and Entrapment Scale (SDES) | Visits 2-5 (24 hours)
  Changes in defeat and entrapment between pre-stimulation (visit 2 and visit 4) and post-stimulation (visit 3 and visit 5), between- and within-person comparisons. The SDES is an 8-item scale measuring defeat and entrapment with 4 items each. Scores range from 0 to 16 per facet (i.e., defeat/entrapment) with higher scores indicating higher defeat and entrapment, respectively.
Beck Depression Inventory (BDI-II) | Visits 2-5 (24 hours)
  Changes in depressive symptoms between pre-stimulation (visit 2 and visit 4) and post-stimulation (visit 3 and visit 5), between- and within-person comparisons. The BDI is a 21-item scale measuring depressive symptoms. Sum scores range from 0 to 63 with higher scores indicating higher severity of depressive symptoms.
Montgomery-Asberg Depression Rating Scale (MADRS) | Visits 2-5 (24 hours)
  Changes in depressive symptoms between pre-stimulation (visit 2 and visit 4) and post-stimulation (visit 3 and visit 5), between- and within-person comparisons. The MADRS is a10-item clinician rating scale measuring depressive symptoms. Scores range from 0 to 60 with higher scores indicating higher severity of depressive symptoms.

OTHER OUTCOMES:
EEG alpha power | Visits 2 & 4 (up to 1 hour)
  Changes in EEG alpha power between pre- and post-stimulation at visit 2 (stimulation visit 1) and visit 4 (stimulation visit 2), between- and within-person comparisons.
EEG: Individual alpha peak frequency | Visits 2 & 4 (up to 1 hour)
  Changes in individual alpha peak frequency between pre- and post-stimulation at visit 2 (stimulation visit 1) and visit 4 (stimulation visit 2), between- and within-person comparisons.
Beck Hopelessness Scale (BHS) | Visits 2-5 (24 hours)
  Changes in hopelessness between pre-stimulation (visit 2 and visit 4) and post-stimulation (visit 3 and visit 5), between- and within-person comparisons. The BHS is a 20-item scale measuring hopelessness. Scores range from 0 to 20 with higher scores indicating increased hopelessness
Perceived Burdensomeness Visual Analogue Scale (PB-VAS) | Visits 2-5 (24 hours)
  Changes in perceived burdensomeness between pre-stimulation (visit 2 and visit 4) and post-stimulation (visit 3 and visit 5), between- and within-person comparisons. The PB-VAS is a single-item visual analogue scale with the statement "I feel like a burden" where 0 indicates "not at all" and 100 indicates "extremely".
Perceived Burdensomeness Visual Analogue Scale (PB-VAS) | Visits 2 & 4 (up to 1 hour)
  Changes in perceived burdensomeness between pre-stimulation at visit 2 and visit 4 and post-stimulation at visit 2 and visit 4, between- and within-person comparisons. The PB-VAS is a single-item visual analogue scale with the statement "I feel like a burden" where 0 indicates "not at all" and 100 indicates "extremely".
Positive and Negative Affective Schedule (PANAS) | Visits 2-5 (24 hours)
  Changes in positive and negative affect between pre-stimulation (visit 2 and visit 4) and post-stimulation (visit 3 and visit 5), between- and within-person comparisons. The PANAS is a 20-item scale measuring positive and negative affect with 10 items each. Scores range from 10 to 50 per domain (i.e. positive & negative affect) where higher scores indicate higher positive or negative affect, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Olbrich, Prof. Dr. med., Principal Investigator — Department of Adult Psychiatry and Psychotherapy, University Hospital of Psychiatry Zurich, University of Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No
Due to ethical considerations and to protect the privacy of study participants, access to data will only be granted following justified requests for research purposes. Deidentified participant data and a data dictionary will then be made available to the requesting person or institution.

REFERENCES:
- [Background] Bankwitz A, Ruesch A, Adank A, Hormann C, Villar de Araujo T, Schoretsanitis G, Kleim B, Olbrich S. EEG source functional connectivity in patients after a recent suicide attempt. Clin Neurophysiol. 2023 Oct;154:60-69. doi: 10.1016/j.clinph.2023.06.025. Epub 2023 Jul 22. PMID 37562347
- See also: OSF Preregistration — https://doi.org/10.17605/OSF.IO/B42J6